CLINICAL TRIAL: NCT05381753
Title: A National Multicenter, Noninterventional Clinical Study Evaluating the Safety and Efficacy of Avapritinib in Chinese Patients With Gastrointestinal Stromal Tumor (GIST) in the Real World
Brief Title: Safety and Efficacy of Avapritinib in Chinese Patients With Gastrointestinal Stromal Tumor (GIST) in the Real World
Status: Completed | Type: Observational
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Avapritinib-4-001
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-11

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; Avapritinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — avapritinib; Imatinib Mesylate; Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (4):
- Ava-mGSIT-P18: Unresectable or metastatic PDGFRA exon 18 GIST
  Interventions: Drug: Avapritinib
- Ava-Perioperative: Perioperative PDGFRA exon 18 GIST
  Interventions: Drug: Avapritinib
- Ava-mGIST-other: Unresectable or metastatic GIST without KIT exon 13，14，or PDGFRA exon 18 mutation
  Interventions: Drug: Avapritinib
- TKI: Unresectable or metastatic PDGFRA exon 18 GIST
  Interventions: Drug: Tyrosine kinase inhibitors other than avapritinib ( imatinib, sunitinib, et al )

INTERVENTIONS:
Drug: Avapritinib — Avapritinib will be administered orally at the starting of 300 mg once daily as the label recommended. Investigators can adjust the dosage, frequency, and duration as needed.
  Groups: Ava-Perioperative; Ava-mGIST-other; Ava-mGSIT-P18
Drug: Tyrosine kinase inhibitors other than avapritinib ( imatinib, sunitinib, et al ) — Investigators will decide which TKI to use as well as the dosage, frequency, and duration.
  Groups: TKI

SUMMARY:
This study is an observational, multicenter, Real-word study to evaluate the safety and clinical efficacy of avapritinib in Chinese subjects with GIST.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 and 4: Participants must have a confirmed diagnosis of unresectable GIST with mutations in the PDGFRα gene exon 18.
* Cohort 2: Participants must have a confirmed diagnosis of GIST with mutations in the PDGFRα gene exon 18 and was/will be administrated avapritinib in an neoadjuvant and/or adjuvant setting.
* Cohort 3: Participants must have a confirmed diagnosis of unresectable GIST without mutations in the PDGFRα gene exon 18, KIT gene exon 13, and KIT gene exon 14.

Exclusion Criteria:

* Participants who have participated and may participate in any other interventional clinical trail in the future.
* Participants with any comorbidities not suitable for avapritinib (other TKIs, Cohort 4) treatment assessed by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GIST patients with specific genetic mutations who were treated or will be treated with avapritinib (other TKIs in corhort 4) in about 20 hospitals from 1 May 2021 to 31 Aug. 2023.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events(AE) and serious adverse events(SAE)in cohort 1, 2, and 3 | AEs were collected from the start of study drug until 30 days after the last dose, SAEs were collected from the date of the informed consent signature until 30 days after the last dose of study drug, up to 3 years.
Dose adjustment of avapritinib in cohort 1, 2, and 3 | From the start of study drug until 30 days after the last dose, up to 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China